CLINICAL TRIAL: NCT02770885
Title: Effects of GLP-1 Analogues on Fluid Intake in Patients With Primary Polydipsia: "The GOLD-Study"
Brief Title: Effects of GLP-1 Analogues on Fluid Intake in Patients With Primary Polydipsia (The GOLD-Study)
Acronym: GOLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOLD 2016
Record Dates: First submitted 2016-03-30; First posted 2016-05-12 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Primary Polydipsia
MeSH Terms: conditions — Polydipsia, Psychogenic | interventions — dulaglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum first (Experimental): Dulaglutide (Trulicity®) 1.5 mg in 0.5 ml, via Pen s.c. once weekly for 3 weeks.
  Interventions: Drug: Dulaglutide
- Placebo first (Placebo Comparator): Placebo: 0.5 ml normal saline (0.9% sodium chloride [0.9% sodium chloride (NaCl)]), injection sc via syringe once weekly for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Treatment with dulaglutide for 3 weeks.
  Other Names: Trulicity
  Arms: Verum first
Drug: Placebo — Treatment with Sodium Chloride 0.9% (Placebo) for 3 weeks.
  Other Names: Sodium Chloride 0.9%
  Arms: Placebo first

SUMMARY:
Glucagon like Peptide -1 (GLP-1) receptor agonists are well known to stimulate glucose-induced insulin secretion and to reduce energy intake. Recent findings from animal and human studies suggest a role of GLP-1 in regulating water and salt homeostasis. GLP-1 has been shown to reduce fluid intake after an oral salt load or during a meal - pointing to a hypodipsic effect. The aim of this study is to elucidate whether these putative hypodipsic properties of GLP-1 might be of advantage in persons with an exaggerated thirst perception as is the case in patients with primary polydipsia.

DETAILED DESCRIPTION:
GLP-1 analogues are currently used for the treatment of hyperglycaemia associated with type 2 diabetes mellitus and given his properties as a natural satiety hormone, the GLP-1 analogue liraglutide was recently approved by the FDA for weight management.

In studies related to the influence of GLP-1 and -analogues in controlling food intake a concomitant reduction of fluid consumption has been observed.

The investigators hypothesize that GLP-1 analogues not only modulate appetite and provide satiety but also reduce fluid intake and thirst sensation in humans - especially in those with excessive thirst perception (patients with primary polydipsia). In view of future therapeutic options for these patients we aim to investigate the influence of the long-acting GLP-1 analogue dulaglutide on fluid intake, thirst perception and quality of life in patients with primary polydipsia compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Polyuria of > 50 ml/Kg/day
* Polydipsia of > 3 liters/day

Exclusion Criteria:

* Known or probable central or nephrogenic Diabetes insipidus, expected from patient's history
* Polyuria secondary to diabetes mellitus, hypokalemia, hypercalcemia
* Pregnancy
* Previous treatment with GLP-1 agonists within the last 3 month
* History of pancreatitis
* Severe renal insufficiency (eGFR (CKD EPI) <30 ml/min/1,73 m2)
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05-17 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Fluid intake in ml | 8 hours
  Fluid intake (ml) during an evaluation visit of 8 hours

SECONDARY OUTCOMES:
Quality of Life Assessment using the Short Form-12 (SF-12) Questionnaire | During phase a and b, 3 weeks each
  To assess the influence of dulaglutide on thirst perception and quality of life in patients with primary polydipsia compared to placebo.
24h-urine production | 24 hours
  24h-urine production in ml during evaluation visit and thereafter
Plasma- and urine osmolality | change during evaluation visit of 8 hours
  influence of dulaglutide on osmolality during evaluation visit
Circadian serum- and salivary cortisol levels | circadian rhythm assessed at timepoints 8am, 12am, 4pm, 8pm and 12pm
  Influence of dulaglutide on hypothalamic-pituitary-adrenal axis (HPA axis) activity
Cortisol levels basal and stimulated | Cortisol at timepoint 0 and after 20-30 minutes after synacthen injection
  Influence of dulaglutide on hypothalamic-pituitary-adrenal axis (HPA axis) activity
Copeptin level | at begin of evaluation 1 day visit after an overnight fast (no drink, no food)
  Influence of dulaglutide on copeptin levels after a period of water deprivation
Influence of dulaglutide on neuronal changes | during phase a and b, 3rd week each for 15 patients
  Neuronal changes assessed with a functional magnet resonance Imaging between dulaglutide and Placebo Treatment in a subgroup of patients with primary polydipsia
Neuronal changes between patients with primary polydipsia and healthy volunteers | for patients during phase a and b, 3rd week each for 15 patients, 15 matched healthy control subjects
  Differences in neuronal changes assessed by functional magnet resonance imaging
Thirst perception | during phase a and b, 3 weeks each and change during evaluation visit of 8 hours
  Influence of dulaglutide on thirst perception

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof, Principal Investigator — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vukajlovic T, Sailer CO, Asmar A, Jensen BL, Vogt DR, Christ-Crain M, Winzeler B. Effect of a 3-Week Treatment with GLP-1 Receptor Agonists on Vasoactive Hormones in Euvolemic Participants. J Clin Endocrinol Metab. 2022 May 17;107(6):e2581-e2589. doi: 10.1210/clinem/dgac063. PMID 35134170
- [Derived] Winzeler B, Sailer CO, Coynel D, Zanchi D, Vogt DR, Urwyler SA, Refardt J, Christ-Crain M. A randomized controlled trial of the GLP-1 receptor agonist dulaglutide in primary polydipsia. J Clin Invest. 2021 Oct 15;131(20):e151800. doi: 10.1172/JCI151800. PMID 34473645